CLINICAL TRIAL: NCT00566657
Title: A Randomized Double-Blind Placebo-Controlled Parallel Group Study of the Efficacy and Safety of XRP0038/NV1FGF on Amputation or Any Death in Critical Limb Ischemia Patients With Skin Lesions
Brief Title: Efficacy and Safety of XRP0038/NV1FGF in Critical Limb Ischemia Patients With Skin Lesions
Acronym: TAMARIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6145; 2006-006277-24 (EudraCT Number)
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: Peripheral Vascular Diseases
Keywords: Critical Limb Ischemia; Peripheral Artery Disease; Plasmid based gene therapy
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease | interventions — riferminogene pecaplasmide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Riferminogene pecaplasmid (Experimental): 4 administrations of riferminogene pecaplasmid 4 mg at 2-week intervals
  Interventions: Biological: riferminogene pecaplasmid
- Placebo (Placebo Comparator): 4 administrations of placebo (for riferminogene pecaplasmid) at 2-week intervals
  Interventions: Biological: Placebo (for riferminogene pecaplasmid)

INTERVENTIONS:
Biological: riferminogene pecaplasmid — Formulation: 5 ml glass vials containing 2,5 ml riferminogene pecaplasmid
  Route: intramuscular (IM) injection of 2.5 mL in the ischemic leg to be treated
  Other Names: NV1FGF; XRP0038
  Arms: Riferminogene pecaplasmid
Biological: Placebo (for riferminogene pecaplasmid) — Formulation: 5 ml glass vials containing 2,5 ml placebo
  Route: IM injection of 2.5 mL in the ischemic leg to be treated
  Arms: Placebo

SUMMARY:
Primary objective is to demonstrate the superiority of riferminogene pecaplasmid (XRP0038/NV1FGF) over placebo in the prevention of major amputation above the ankle of the treated leg or of death from any cause, whichever comes first, in critical limb ischemia (CLI) patients with skin lesions.

Secondary objectives are to evaluate:

* The efficacy of riferminogene pecaplasmid versus placebo for delaying the time to major amputation;
* The efficacy of riferminogene pecaplasmid versus placebo for delaying the time to death;
* The safety of riferminogene pecaplasmid in the study population.

DETAILED DESCRIPTION:
The study consists in 6-week treatment then a follow-up period up to 12 months. A follow-up contact is then scheduled 6 months later.

Per protocol amendment a 18-month long-term safety survey was added.

ELIGIBILITY:
Inclusion Criteria:

* Having peripheral artery disease at the stage of Critical Limb Ischemia (CLI) with skin lesions (either ulcer(s) or gangrene);
* With objective evidence of CLI such as ankle systolic pressure <70 mmHg and/or toe systolic pressure <50 mmHg or transcutaneous oxygen pressure (TcPO2) <30 mmHg;
* Unsuitable for standard revascularization of his/her peripheral arterial disease;
* Having a negative screening for cancer.

Exclusion Criteria:

* Previous major amputation on the leg to be treated or planned major amputation within the first month following randomization;
* Known Buerger's disease;
* Successful lower extremity revascularization procedure within 3 months prior randomization;
* Uncontrolled blood pressure defined as systolic blood pressure (SBP) ≥180 mmHg or diastolic blood pressure (DBP) ≥110 mmHg despite adequate antihypertensive treatment;
* Acute cardiovascular events within 3 months prior to randomization;
* Active proliferative retinopathy and severe macular oedema;
* Previous or current history of malignant disease within the past 5 years;
* Previous treatment with systemic angiogenic factors or with stem cells therapy;
* Pregnant or breast-feeding woman or woman of childbearing potential not protected by an effective contraceptive method of birth control. Man not following effective contraceptive method with his partner of childbearing potential during the course of the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2007-11; Primary Completion 2010-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Time to major amputation of the treated leg or death from any cause, whichever comes first | From randomization up to 12 months

SECONDARY OUTCOMES:
Time to first major amputation of the treated leg | From randomization up to 12 months
Time to death from any cause | From randomization up to 12 months
Number of participants with adverse events as a measure of safety | From 1st treatment administration up to death, or the earliest of Day 360 or last contact/assessment

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (32):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Minsk, Belarus
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Tatari, Estonia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Tokyo, Japan
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Kiev, Ukraine
- Sanofi-Aventis Administrative Office, Guildford, Surrey, United Kingdom

REFERENCES:
- [Result] Van Belle E, Nikol S, Norgren L, Baumgartner I, Driver V, Hiatt WR, Belch J. Insights on the role of diabetes and geographic variation in patients with critical limb ischaemia. Eur J Vasc Endovasc Surg. 2011 Sep;42(3):365-73. doi: 10.1016/j.ejvs.2011.04.030. Epub 2011 Jun 21. PMID 21696982
- [Result] Belch J, Hiatt WR, Baumgartner I, Driver IV, Nikol S, Norgren L, Van Belle E; TAMARIS Committees and Investigators. Effect of fibroblast growth factor NV1FGF on amputation and death: a randomised placebo-controlled trial of gene therapy in critical limb ischaemia. Lancet. 2011 Jun 4;377(9781):1929-37. doi: 10.1016/S0140-6736(11)60394-2. Epub 2011 May 28. PMID 21621834